CLINICAL TRIAL: NCT06061068
Title: The Effect of Hernia Belt on Postoperative Complications and Quality of Life for Patients Who Underwent Laparoscopic Inguinal Hernia Repair:a Randomized Clinical Trial
Brief Title: Hernia Belt in Laparoscopic Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Collaborators: Guang'an People's Hospital (Unknown); Pengan County People's Hospital (Other); People's Hospital of Yilong County (Unknown); Nanbu Hospital of County Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yunhong Tian, Director of Gastrointestinal, Colorectal and Hernia Surgery, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230910
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hernia, Inguinal; Recurrence; Seroma Following Procedure; Pain, Postoperative; Quality of Life
Keywords: Laparoscopic inguinal hernia repair; Hernia belt; Hernia recurrence; Seroma Following Procedure; Pain, Postoperative; Quality of Life
MeSH Terms: conditions — Hernia, Inguinal; Recurrence; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hernia belt compressing group (Experimental): Patients were given hernia belt compression of the inguinal region after laparoscopic inguinal hernia repair surgery in the operating room. The silicone pad of the hernia belt was placed in the inguinal region of the surgical side for compression for a period of 2 weeks.
  Interventions: Procedure: Hernia belt compression
- No hernia belt compressing group (No Intervention): Patients were should not have the intervention "Hernia belt compression" .

INTERVENTIONS:
Procedure: Hernia belt compression — Use the hernia belt to compress the inguinal region
  Arms: Hernia belt compressing group

SUMMARY:
In this study, the investigators aimed to investigate the effect of hernia belt on postoperative complications and quality of life for patients who underwent laparoscopic inguinal hernia repair. Outcomes include hernia recurrence (patient-reported and clinical exam), postoperative complications within 3 months (seroma and hematoma development, wound infection, abdominal bloating and foreign body sensation), pain (visual analog scale,VAS), health-related quality of life (36-item short-form health survey, SF-36). Follow up by physical examination, ultrasonography and telephone.

DETAILED DESCRIPTION:
Some scholars believe that the use of hernia belts to compress the inguinal region reduces postoperative complications. According to the International Guidelines for the Management of Inguinal Hernia in Adults (2018) interpretation, the incidence of seroma after inguinal hernia repair ranges from 0.5% to 2.2%. However,there is no consensus among different research organizations and clinical staff on the use of hernia belts after laparoscopic inguinal hernia repair. In this study, the investigators aimed to investigate the effect of hernia belt on postoperative complications and quality of life for patients who underwent laparoscopic inguinal hernia repair. Outcomes include hernia recurrence (patient-reported and clinical exam), postoperative complications within 3 months (seroma and hematoma development, wound infection, abdominal bloating and foreign body sensation), pain (visual analog scale,VAS), health-related quality of life (36-item short-form health survey, SF-36). Follow up by physical examination, ultrasonography and telephone.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or order.
2. Primary unilateral oblique inguinal hernia, direct hernia, femoral hernia.
3. Qualified for laparoscopic Transabdominal preperitoneal approach(TAPP) or Totally extraperitoneal(TEP).
4. Eligible to tolerate general anesthesia.

Exclusion Criteria:

1. Incarcerated hernia, recurrent hernia and other types of hernia.
2. Patients presenting for obvious contraindications to surgery.
3. Need for an open inguinal hernia repair.
4. Difficult to follow-up or communication.
5. Patients who are unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 1 month,3 months,6 months and 12 months after surgery.
  Follow up by physical examination, ultrasonography and telephone at 1 month,3 months,6 months and 12 months after surgery about the rate of hernia recurrence.
Postoperative complications | Within 3 months after surgery.
  Including seroma and hematoma development, wound infection, abdominal bloating and foreign body sensation,follow up by physical examination, ultrasonography and telephone.
Pain score | 1 day,7 days,1 month and 3 months after surgery.
  The visual analog scale (VAS) was adopted for pain evaluation preoperative,1 day, 7 days, 1 months and 3 months postoperatively.The scale range from 0 to 10, with 0 meaning no pain and 10 meaning the worst pain.Higher scores mean a worse outcome.
Health-related quality of life | 1 day,7 days,1 month and 3 months after surgery.
  The 36-item short-form health survey(SF-36) was adopted for Health-related quality of life 1 day, 7 days, 1 months and 3 months postoperatively. SF-36 consists of 36 articles, including 8 areas of physical function, physical role, physical pain, general health status, vitality, social function, emotional role and mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China